CLINICAL TRIAL: NCT06795711
Title: Validation and Optimisation of Ultrasound Diagnosis of Adenomyosis: a Prospective Observational Study
Brief Title: Validation and Optimisation of Ultrasound Diagnosis of Adenomyosis
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ADENAS
Record Dates: First submitted 2024-12-03; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-11

CONDITIONS: Adenomyosis
Keywords: adenomyosis; gynaecology; ultrasound
MeSH Terms: conditions — Adenomyosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Defining ultrasound criteria for normal uterine biometry and assessing the prevalence of repeat abortions in patients with abnormalities of the uterine cavity

DETAILED DESCRIPTION:
Adenomyosis is a gynaecological disorder with a high prevalence in women of childbearing age and is characterised by the presence of glands and endometrial stroma within the myometrium, associated or not with hypertrophy and hyperplasia of the surrounding myometrium. Adenomyosis may cause pelvic pain and/or abnormal uterine bleeding. Transvaginal ultrasound may be considered the main non-invasive diagnostic modality for the diagnosis of adenomyosis. The aim is to optimise the ultrasound diagnosis of uterine pathology and in particular of adenomyosis by defining uterine biometric parameters (longitudinal, transverse and anteroposterior diameters and their ratios; uterine volume) allowing patients to be divided into 3 groups:

* Uterus affected by adenomyosis (group A): adenomyosis is a gynaecological condition with high prevalence in women of childbearing age and is characterised by the presence of endometrial tissue (innermost layer of the uterus) within the uterine muscle. Adenomyosis can cause abdominal pain and abnormal uterine bleeding.
* Uterus affected by fibromatosis (group B): uterine fibromatosis is a gynaecological condition characterised by the appearance of numerous fibroids in the uterus. It is a very frequent condition in the general population and its frequency increases as the age of the patients increases.
* Normal uterus (group C). Transvaginal ultrasound, although a reference diagnostic tool, still remains an operator-dependent examination to date: our secondary objective is to build models that can simplify diagnosis through the use of artificial intelligence. The aim is to create various artificial intelligence software that can 'learn to make a diagnosis'. This method has already been applied in radiology, proving capable of discriminating between benign and malignant tumours from images from different diagnostic methods with performance similar to that of experienced radiologists.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 60;
* obtaining informed consent

Exclusion Criteria:

* Hysterectomised patients;
* Virgo patients (hymenal integrity);
* Patients reporting intolerance to transvaginal ultrasound;
* Gynaecological oncology;
* Recent pregnancy or childbirth (within 6 months);
* Menopausal patients

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients consecutively attending our ultrasound clinics for routine check-ups or pre-operative examinations will be included, as per regular practice. For the purposes of the analysis, patients will be divided into three groups according to the ultrasound and/or surgical diagnosis of A adenomyosis (presence of at least 2 ultrasound signs compatible with adenomyosis (MUSA) or presence of glands and endometrial stroma in myometrial location), B fibromatosis (uterus with inhomogeneous echostructure lacking 2 or more signs compatible with uterine adenomyosis or histological finding of several benign tumours consisting of smooth muscle tissue and fibrous tissue in varying proportions), C normal uterus (normal echostructure on transvaginal ultrasound)
Sampling Method: Non-Probability Sample
Enrollment: 465 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Definition of uterine biometric parameters | After enrollment on first visit
  Definition of uterine biometric parameters for the diagnosis of adenomyotic uterus (group A), fibromatous uterus (group B) and normal uterus (group C) by means of transvaginal ultrasound, performed as per the care procedure. Evaluation of the diagnostic capacity of 'globular uterus' for the diagnosis of adenomyosis as an additional parameter to those already known in the literature with possible subsequent identification of a biometric cut-off
Diagnostic capacity of 'globular uterus' for the diagnosis of adenomyosis | After enrollment on first visit
  Evaluation of the diagnostic capacity of 'globular uterus' for the diagnosis of adenomyosis as an additional parameter to those already known in the literature with possible subsequent identification of a biometric cut-off

SECONDARY OUTCOMES:
Construction of deep learning models on uterine ultrasound images | After enrollment on first visit
  Construction of deep learning models trained, validated and tested on uterine ultrasound images for the ultrasound diagnosis of adenomyosis and evaluation of their diagnostic accuracy
Evaluation of diagnostic accuracy of deep learning validated | After enrollment on first visit
  Evaluation of diagnostic accuracy of deep learning validated for ultrasound diagnosis of adenomyosis
Identification of the frequency of finding ultrasound signs of adenomyosis in the cervix | After enrollment on first visit
  In patients with a diagnosis of adenomyosis made on the basis of ultrasound features at the level of the uterine body and fundus
Evaluation of diagnostic accuracy | After enrollment on first visit
  Evaluation of the diagnostic accuracy of trainees when experienced (identifying experienced operators as doctors in specialised training in Gynaecology and Obstetrics for at least four years, with an experience of at least 500 gynaecological ultrasound cases) and moderately experienced (identifying moderately experienced operators as doctors in specialised training in Gynaecology and Obstetrics for at least two years, with an experience of at least 200 gynaecological ultrasound cases

CONTACTS AND LOCATIONS:
Overall Officials: Diego Raimondo, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy